CLINICAL TRIAL: NCT01751633
Title: Comparison of Surgical Versus Conservative Treatment of AO Type A3 Thoracolumbar Fractures Without Neurological Deficits Prospective, International, Multicenter Cohort Study
Brief Title: Spine FA3 - a Prospective, International, Multicenter Cohort Study on Treatment of of AO A3 Thoracolumbar Fractures
Acronym: FA3
Status: Terminated | Type: Observational
Why Stopped: Administrative reason. Lack of funding.
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: Spine FA3
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Single Level Stable Thoracolumbar Fracture Type AO A3; Multiple Level Stable Thoracolumbar Fracture Type AO A3
Keywords: Burst fractures; Thoracic or Lumbar Vertebrae/injuries [MeSH]; Thoracic or Lumbar Vertebrae/surgery [MeSH]; Spinal Fusion/methods [MeSH]; Thoracolumbar fracture management; Quality of life; Functional outcome
MeSH Terms: interventions — Surgical Procedures, Operative; Conservative Treatment; Calcium Sulfate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surgical treatment: Surgical treatment according to one of the following:
  * Posterior open approach
  * Posterior minimally-invasive surgery (MIS) approach The choice of the approach will be left upon the surgeon's discretion
  Interventions: Procedure: Surgical
- Conservative treatment: Conservative treatment according to hospital's standard of care
  Interventions: Procedure: Conservative treatment

INTERVENTIONS:
Procedure: Surgical
  Other Names: • Posterior open approach; • Posterior minimally-invasive surgery (MIS) approach
  Groups: Surgical treatment
Procedure: Conservative treatment
  Other Names: Conservative treatment according to hospital's standard of care :; - Bed rest followed by immobilization with:; - Custom-moulded or prefabricated total body contact thoracolumbosacral orthosis (TLSO); - Thermoplastic removable brace, Jewett hyperextension braces, Anterior hyperextension brace (ASH), Taylor-Knight brace; - Plaster of Paris (POP)
  Groups: Conservative treatment

SUMMARY:
Thoracolumbar fractures are the most common spinal fractures with an average annual incidence between 18 and 30 per 100'000 inhabitants. The majority of these fractures are AO type A3 ("burst fractures"). Although patients with burst fractures report a reduced quality of life and chronic pain, there is no clear evidence whether surgical or conservative treatment offer better functional and back-pain related outcomes. The indications for the selection of an ideal treatment for these fractures without neurological deficits remain controversial. The purpose of this study is to evaluate whether patients with thoracolumbar fractures without neurological deficit being surgically treated show faster recovery and better improvement of function than patients being conservatively treated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Diagnosis of single or multiple stable thoracolumbar fracture(s)

  * Level T10- L3
  * Type AO A3 or A4
  * Radiologically confirmed by Rx or CT
* Fracture induced kyphotic deformity lower or equal to 20-35 degrees
* Definitive treatment (surgical or conservative) within 10 days after injury
* American Spinal Injury Association (ASIA) Impairment Scale = E (normal )
* Ability to understand patient information / informed consent form
* Willingness and ability to participate in the clinical investigation including imaging and follow-up procedures (FUs)
* Signed informed consent

Exclusion Criteria:

* Open fracture
* Polytrauma
* Pathologic fracture
* Disruption of the posterior ligamentous complex between T10 and L3
* Clinically evident osteoporosis as assessed by the investigator
* Spinal luxation
* Associated severe lesions as assessed by the investigator
* Spinal lesion due to gun or projectile
* Pre-existing spinal column deformity
* Prior spinal surgeries
* BMI > 40 kg/m2
* Any severe medically not managed systemic disease
* Recent history of substance abuse (ie, recreational drugs, alcohol) that would preclude reli-able assessment
* Pregnancy or women planning to conceive within the study period
* Prisoner
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 140 subjects patients with thoracolumbar fractures will be assigned to ei-ther conservative or surgical treatment depending on the surgeon's decision. Patients will be treated at each institution per standard of care. Surgeons will use their expertise and preferences to determine the method of surgical or conservative intervention.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Roland-Morris Disability Questionnaire (RMDQ) | 6 week follow up
  Improvement in functional outcome from baseline to 6 week follow up (FU) measured with the Roland-Morris Disability Questionnaire (RMDQ)

SECONDARY OUTCOMES:
Back pain related disability (Roland-Morris Disability Questionnaire RMDQ) | Assessed at baseline, 6 weeks, 3, 6, 12 and 24 months follow up
Pain (Numeric Rating Scale (NRS)) | Assessed at baseline, 6 weeks, 3, 6, 12 and 24 months FU
Radiologic progress taking into account RX, CT and optionally MRI | baseline and at follow up after 6 weeks, 3, 6, 12 and 24 months
Quality of return to work (Denis Work Scale) | Assessed at baseline, 6 weeks, 3, 6, 12 and 24 months follow up
Time to return to work | Assessed at baseline, 6 weeks, 3, 6, 12 and 24 months follow up
Conservative treatment failure rate (eg, change to surgical treatment) | Assessed at baseline, 6 weeks, 3, 6, 12 and 24 months follow up
Rates of local adverse events (AE) | Assessed at baseline, 6 weeks, 3, 6, 12 and 24 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Barbagallo, MD, Principal Investigator — Azienda Ospedaliero - Universitaria Policlinico, Catania, Italy; Emiliano Vialle, MD, Principal Investigator — Catholic University of Parana - Curitiba, Brazil
Locations (8):
- Brazil (3):
  - Hospital Universitaria Cajuru, Curitiba
  - Hospital Cristo Redentor, Porto Alegre
  - Hospital Santa Marcelina, São Paulo
- Hospital Cristo Redentor, Santiago, Chile
- Krajská nemocnice Liberec, Liberec, Czechia
- Klinikum rechts der Isar der Technischen Universität München, Munich, Germany
- Azienda Ospedaliero - Universitaria Policlinico, Catania, Italy
- Hospital Garcia e Orta, EPE, Almada, Portugal